CLINICAL TRIAL: NCT01391598
Title: Evaluation of the Effect of Intravenous Lidocaine on Pain Relief and Plasma Concentrations of Interleukins (IL-1 and IL-6) and Substance P in Patients With Fibromyalgia
Brief Title: Lidocaine on Pain Relief and IL and Substance P in Fibromyalgia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Ana Laura Albertoni Giraldes, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FibromialgiaGiraldes
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2009-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; intravenous lidocaine; substance P; interleukins
MeSH Terms: conditions — Fibromyalgia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): After completion of the inclusion criteria all patients receive a dose of amitriptyline 12.5 mg in the first week, and 25 mg in the eight subsequent weeks, orally, once daily at night. At lidocaine group 20 pacients will receive lidocaine at a dose of 4 mg / kg, not exceeding a dose of 240 mg diluted in 125ml of solution 0.9% saline.The solutions will be infused in 1 hour once a week in the four weeks following the start of the study..:Patients may use as additional analgesics up to 4g/day acetaminophen, and if necessary, they can use tramadol, recording the dose
  Interventions: Drug: Lidocaine
- Saline (Placebo Comparator): After completion of the inclusion criteria all patients receive a dose of amitriptyline 12.5 mg in the first week, and 25 mg in the eight subsequent weeks, orally, once daily at night. At saline group 20 pacients will receive 125ml of solution 0.9% saline.The solutions will be infused in 1 hour once a week in the four weeks following the start of the study. Patients may use as additional analgesics up to 4g/day acetaminophen, and if necessary, they can use tramadol, recording the dose
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: Lidocaine — After completion of the inclusion criteria all patients receive a dose of amitriptyline 12.5 mg in the first week, and 25 mg in the eight subsequent weeks, orally, once daily at night. At lidocaine group 20 pacients will receive lidocaine at a dose of 4 mg / kg, not exceeding a dose of 240 mg diluted in 125ml of solution 0.9% saline.The solutions will be infused in 1 hour once a week in the four weeks following the start of the study..:Patients may use as additional analgesics up to 4g/day acetaminophen, and if necessary, they can use tramadol, recording the dose
  Arms: Lidocaine
Drug: lidocaine — After completion of the inclusion criteria all patients receive a dose of amitriptyline 12.5 mg in the first week, and 25 mg in the eight subsequent weeks, orally, once daily at night. At saline group 20 pacients will receive 125ml of solution 0.9% saline.The solutions will be infused in 1 hour once a week in the four weeks following the start of the study. Patients may use as additional analgesics up to 4g/day acetaminophen, and if necessary, they can use tramadol, recording the dose
  Arms: Saline

SUMMARY:
The study's primary objective is to evaluate the effect of intravenous lidocaine on pain and plasma interleukin-1 (IL-1), interleukin-6 (IL-6) and substance P in patients with fibromyalgia.

As secondary objectives: evaluate the clinical manifestations, and plasma concentration of lidocaine.

DETAILED DESCRIPTION:
Fibromyalgia is a painful syndrome characterized by chronic diffuse pain and involvement of multiple muscles and soft tissues 1. The pain is very common, with prevalence around 2% in the adult population.

In fibromyalgia, there is an increase of both somatic and visceral nociception, and dysfunction of central nervous.system According to the American College of Rheumathology diagnostic criteria for fibromyalgia are widespread pain and the presence of 11 of 18 typical tender points 3.

Minor criteria in the inclusion of patients for the diagnosis of fibromyalgia, such as pain that changes with physical activity, sleep disturbance, fatigue, anxiety, depression, paresthesia, cramps, sensation of swelling 4. Several co-morbidities may be associated with pain such as migraine, myofascial pain syndrome, and irritable bowel syndrome.

The symmetry of these conditions shows that fibromyalgia is associated with central sensitization 5. The pathophysiological mechanisms of fibromyalgia are related to changes in neurotransmitters 6,7,8. Cytokines may be involved in modulation of symptoms such as hyperalgesia, fatigue and depression, and maintenance of sympathetic pain 9.

] The substance P ( SP ) levels are increased in cerebrospinal fluid of patients with fibromyalgia compared to control groups 10.

Antidepressants are the most widely used drugs for its treatment. The drug most commonly used is amitriptyline.

Other drugs (muscle relaxants, anticonvulsants, NSAIDs, tramadol) are also employed. Physical activity is essential to control the symptoms. Physical measures, psychotherapy, occupational therapy are other treatments, but the effectiveness is variable 14.15. Sometimes a combination of drugs and techniques are needed to obtain satisfactory results.

The infusion of local anesthetic is given intravenously for fibromyalgia when oral medication does not produce the proper effect. It promotes sympathetic blockade, vasodilation, anesthesia of the nerve endings in the vascular endothelium, stabilization of membrane and breaks the vicious circle that keeps pain 16.

Local anesthetics are membrane-stabilizing and prevent the generation of ectopic impulses in lower concentrations than those needed to block the normal driving. The dose used by different authors ranged from 1 to 5 mg / kg, administered in 30-60 minutes 17-24. Side effects of lidocaine are: sedation, vertigo, dizziness, blurred vision, nausea and vomiting 25.

The effectiveness of intravenous lidocaine in neuropathic pain is well established 26. Despite evidence of analgesic effect, there is controversy in conditions without nerve injury. It may be that the selectivity of the effect for non-neuropathic and neuropathic pain is relative and depends on the plasma concentration reached25.

For the use of systemic lidocaine in fibromyalgia, there are no well-controlled studies, and to assess changes of cytokines and substance P, which stimulated this research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fibromyalgia will be included in the study through the classification criteria proposed by the American College of Rheumatology (generalized hypersensitivity and pain or stiffness in 11 of 18 musculotendinous insertions sites for at least three months in the four quadrants of the body, absence of traumatic injury, rheumatic disease, neuromuscular or infectious arthropathy).

Exclusion Criteria:

* Will be excluded from the study patients who had: no cognitive or language comprehension; abnormal laboratory tests, trauma, psychiatric illness, rheumatic or neuromuscular another pain syndrome, infectious arthropathy, hypersensitivity to drugs and pregnant. Also will be excluded patients with arrhythmia, myocardial infarction, concomitant use of cisapride or monoamine oxidase inhibitor, bundle branch block or atrio-ventricular heart failure, acute, angle glaucoma, myasthenia gravis, severe liver disease and hyperthyroidism; and those who are using centrally acting analgesic medication (antidepressants, anticonvulsants, opioids, neuroleptics) for at least 4 weeks from baseline.

Patients who experience severe side effects related to the infusion of lidocaine (severe hypotension and seizure) will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of intravenous lidocaine on pain relief and plasma concentrations of interleukins (IL-1 and IL-6) and substance P in patients with fibromyalgia | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Unifesrity of Sao Paulo, São Paulo, São Paulo, Brazil